CLINICAL TRIAL: NCT06400368
Title: Proof of Concept of the Effect of LEQEMBI on Cerebral and Retinal Amyloid in Mild Cognitive Impairment Due to Alzheimer's Disease
Brief Title: Effect of LEQEMBI on Cerebral and Retinal Amyloid in Mild Cognitive Impairment Due to Alzheimer's Disease
Status: Recruiting | Type: Observational
Sponsor: NeuroVision Imaging (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023.128-1
Record Dates: First submitted 2024-04-29; First posted 2024-05-06 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease
Keywords: retinal image; CAA; Leqembi; lecanamab
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a proof of concept observational study is to determine if there is correlation between Aβ plaques and vascular findings in the Retina versus brain ARIA.

DETAILED DESCRIPTION:
Based upon studies and histological evidence, investigators and study sponsor suspects that the primary mechanism that causes CAA in the brain (and increased risk of ARIA) may also occur in the retina. Investigators propose use of both amyloid brain PET imaging, MRI, and retinal imaging to determine if patients undergoing Lecanemab treatment allows for in the ability to correlate ARIA from retinal amyloid and vasculature versus MRI criteria, and a measurable reduction in amyloid in the retina when compared with amyloid PET scans of the brain post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be eligible for and intend to receive LEQEMBI under standard of care treatment.
2. Male and female subjects ages ≥50 years old.
3. Must be willing to comply with protocol including pupillary dilation to a minimum of 3.5 mm to allow for ocular imaging.
4. Patient or patient's legally authorized representative (LAR) (e.g., spouse or legal guardian) has the ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local patient privacy regulations.

Exclusion Criteria:

1. History of acute angle-closure glaucoma or allergic reaction to the protocol-specified ophthalmic medication for dilation of the pupils.
2. Self-reported or diagnosed history of dense cataracts or other significant media opacity that may affect clear images of the retina.
3. Subjects must not have had eye surgery in the past 2 months, be currently administering eye drops relating to previous eye surgery,
4. Unable or unwilling to comply with the protocol requirements.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female subjects ages 50 and up eligible for treatment with LEQEMBI.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Investigational and Research- retinal vessel and tortuosity | From enrollment to the end of the treatment at 1 year.
  Measurements of amyloid levels in the retina based on autoflourescence imaging, retinal vessel and tortuosity.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Kile, MD, Principal Investigator — Sutter Health
Locations (1):
- Sutter Health, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No